CLINICAL TRIAL: NCT01841450
Title: A Prospective, Controlled, Multicenter Post-Approval Study Of The Glaukos® iStent® Trabecular Micro-Bypass Stent System In Conjunction With Cataract Surgery
Brief Title: Multicenter Post-Approval Study Of The Glaukos® iStent® Trabecular Micro-Bypass Stent System In Conjunction With Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTS100-PAS2 (Rev1 04-11-2016)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open-angle glaucoma (POAG); Trabecular meshwork; iStent
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iStent (Experimental): Implantation of one iStent in conjunction with cataract surgery
  Interventions: Device: iStent
- Cataract surgery (Active Comparator): Cataract surgery alone
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Device: iStent — Implantation of one iStent in conjunction with cataract surgery
  Other Names: GTS100
  Arms: iStent
Procedure: Cataract surgery — Cataract surgery alone
  Arms: Cataract surgery

SUMMARY:
The purpose of this study is to assess the long-term safety of the Glaukos® iStent® Trabecular Micro-Bypass Stent Model GTS100 in conjunction with cataract surgery vs. cataract surgery only, in subjects with mild to moderate open-angle glaucoma.

DETAILED DESCRIPTION:
The purpose of this study is to assess the long-term safety of the Glaukos® iStent® Trabecular Micro-Bypass Stent Model GTS100 in conjunction with cataract surgery compared to cataract surgery only, in subjects with mild to moderate open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate primary open-angle glaucoma
* currently treated with ocular hypotensive medication
* pseudoexfoliative and pigmentary glaucoma are acceptable diagnoses
* subject scheduled to undergo cataract surgery

Exclusion Criteria:

* primary angle-closure glaucoma; or secondary angle closure glaucoma, including neovascular glaucoma
* retrobulbar tumor, thyroid eye disease, Sturge-Weber syndrome or any other type of condition that may cause elevated episcleral venous pressure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Rate of sight-threatening adverse events | 36 months

SECONDARY OUTCOMES:
Other adverse events | 36 months
  For other adverse events such as increase in intra-ocular pressure (IOP) of ≥ 10 mmHg at any time postoperative, loss of best spectacle corrected visual acuity of ≥ 2 lines (≥ 10 letters) postoperative as compared to baseline or best recorded visual acuity measured at any visit postoperative, the rate of each event at each visit will be calculated for the two treatment groups separately.

OTHER OUTCOMES:
Diurnal IOP reduction ≥ 20% | Baseline and 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Irvine, California
  - Montebello, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Jackson, Michigan
  - Saint Joseph, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Mentor, Ohio
  - Kingston, Pennsylvania